CLINICAL TRIAL: NCT05415722
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2a Clinical Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Orally Administered TERN-501 as Monotherapy as Well as in Combination With TERN-101 in Noncirrhotic Adults With Presumed Non-Alcoholic Steatohepatitis (NASH)
Brief Title: DUET Study: A Clinical Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Orally Administered TERN-501 as Monotherapy and in Combination With TERN-101 in Noncirrhotic Adults With Presumed Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Terns, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TERNCB-2002
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic steatohepatitis (NASH); FXR agonist; Nonalcoholic Fatty Liver Disease (NAFLD); THR-β agonist
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1: TERN-501 1 mg (Experimental): Orally administered.
  Interventions: Drug: TERN-501
- Arm 2: TERN-501 3 mg (Experimental): Orally administered.
  Interventions: Drug: TERN-501
- Arm 3: TERN-501 6 mg (Experimental): Orally administered.
  Interventions: Drug: TERN-501
- Arm 4: TERN-501 3 mg + TERN-101 10 mg (Experimental): Orally administered.
  Interventions: Drug: TERN-501; Drug: TERN-101
- Arm 5: TERN-501 6 mg + TERN-101 10 mg (Experimental): Orally administered.
  Interventions: Drug: TERN-501; Drug: TERN-101
- Arm 6:TERN-101 10 mg (Experimental): Orally administered.
  Interventions: Drug: TERN-101
- Arm 7: Matching placebo (Placebo Comparator): Orally administered.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TERN-501 — Investigational drug
  Arms: Arm 1: TERN-501 1 mg; Arm 2: TERN-501 3 mg; Arm 3: TERN-501 6 mg; Arm 4: TERN-501 3 mg + TERN-101 10 mg; Arm 5: TERN-501 6 mg + TERN-101 10 mg
Drug: TERN-101 — Investigational drug
  Arms: Arm 4: TERN-501 3 mg + TERN-101 10 mg; Arm 5: TERN-501 6 mg + TERN-101 10 mg; Arm 6:TERN-101 10 mg
Other: Placebo — Matching placebo
  Arms: Arm 7: Matching placebo

SUMMARY:
This is a Phase 2a Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Orally Administered TERN-501 as Monotherapy as well as in Combination with TERN-101 in Noncirrhotic Adults with Presumed Non-Alcoholic Steatohepatitis (NASH)

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Overweight or obese with a body mass index (BMI) ≥ 25 kg/m2
* Presumed NASH diagnosed by prior biopsy and/or imaging criteria
* Written informed consent

Key Exclusion Criteria:

* History or clinical evidence of chronic liver diseases other than NAFLD
* History or known clinical evidence of cirrhosis, esophageal varices, hepatic decompensation or other severe liver impairment,
* History of liver transplant, or current placement on a liver transplant list
* Current diagnosis or history of pituitary or thyroid disorders - except for patients with primary hypothyroidism on a stable dose of thyroid hormone replacement therapy.
* Abnormal TSH or free T4 levels
* Weight loss of > 5% total body weight within 3 months prior to Screening
* Uncontrolled diabetes
* Uncontrolled hyperlipidemia
* Unstable cardiovascular disease
* Excessive alcohol consumption

Other protocol-defined I/E criteria that apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Terns, Inc.
Locations (35):
- United States (35):
  - Site 1017: The Institute for Liver Health dba Arizona Liver Health, Chandler, Arizona
  - Site 1018: Arizona Liver Health, Tucson, Arizona
  - Site 1004 Southern California Research Center, Coronado, California
  - Site 1061 Velocity Clinical Research, Gardena, Gardena, California
  - Site 1013 University of California, San Diego - Altman Clinical and Translational Research Institute, La Jolla, California
  - Site 1016 Ruane Clinical Research Group Inc., Los Angeles, California
  - Site 1060 Catalina Research Institute, LLC, Montclair, California
  - Site 1001 National Research Institute, Panorama City, California
  - Site 1040 Inland Empire Clinical Trials, LLC, Rialto, California
  - Site 1062 Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Site 1057:Integrity Clinical Research, LLC, Doral, Florida
  - Site 1041: Florida Research Institute, Lakewood Rch, Florida
  - Site 1058 Optimus U Corporation, Miami, Florida
  - Site 1036 Schiff Center for Liver Diseases / University of Miami, Miami, Florida
  - Site 1045 University of Miami Hospital & Clinics, Sylvester Comp. Cancer Center, Miami, Florida
  - Site 1007: Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Site 1055: Progressive Medical Research, Port Orange, Florida
  - Site 1032 IU Health University Hospital, Indianapolis, Indiana
  - Site 1052: Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Site 1054 Louisiana Research Center, Shreveport, Louisiana
  - Site 1063 GI Alliance - Flowood, Flowood, Mississippi
  - Site 1042: Lucas Research, Inc, Morehead City, North Carolina
  - Site 1059: Premier Medical Group, Clarksville, Tennessee
  - Site 1044: Quality Medical Research, Nashville, Tennessee
  - Site 1005:Texas Clinical Research Institute, LLC, Arlington, Texas
  - Site 1050: Pinnacle Clinical Research, Austin, Texas
  - Site 1051: South Texas Research Institute, Edinburg, Texas
  - Site 1043 Liver Specialists of Texas, Houston, Texas
  - Site 1046 Houston Methodist Hospital, Houston, Texas
  - Site 1039: Houston Research Institute, Houston, Texas
  - Site 1003: Clinical Trials of Texas, LLC, San Antonio, Texas
  - Site 1006: American Research Corporation, San Antonio, Texas
  - Site 1056: Pinnacle Clinical Research, San Antonio, Texas
  - Site 1053 Bon Secours Richmond Community Hospital LLC d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Site 1022 Liver Institute Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noureddin M, Alkhouri N, Lawitz EJ, Kowdley KV, Loomba R, Lee L, Jones C, Schlegel A, Marmon T, Anderson K, Li Y, Quirk E, Harrison SA. TERN-501 monotherapy and combination therapy with TERN-101 in metabolic dysfunction-associated steatohepatitis: the randomized phase 2a DUET trial. Nat Med. 2025 Jul;31(7):2297-2305. doi: 10.1038/s41591-025-03722-7. Epub 2025 Jun 11. PMID 40500414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 591 patients were screened with 429 patients failing screening.
Period: Overall Study
Arm/Group | Arm 1: TERN-501 1 mg | Arm 2: TERN-501 3 mg | Arm 3: TERN-501 6 mg | Arm 4: TERN-501 3 mg + TERN-101 10 mg | Arm 5: TERN-501 6 mg + TERN-101 10 mg | Arm 6:TERN-101 10 mg | Arm 7: Matching Placebo
Started | 23 | 23 | 22 | 23 | 23 | 24 | 24
Treated | 23 | 23 | 22 | 23 | 23 | 24 | 24
Discontinued Treatment (Patient completed the study but did not complete the treatment) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Completed (Patient completed the study) | 23 | 20 | 22 | 19 | 21 | 23 | 21
Not Completed | 0 | 3 | 0 | 4 | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Discretion | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients who were randomized and received at least 1 dose of study drug were included in the Efficacy Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: TERN-501 1 mg | Arm 2: TERN-501 3 mg | Arm 3: TERN-501 6 mg | Arm 4: TERN-501 3 mg + TERN-101 10 mg | Arm 5: TERN-501 6 mg + TERN-101 10 mg | Arm 6:TERN-101 10 mg | Arm 7: Matching Placebo | Total
Number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 24 | 24 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 19 | 16 | 20 | 20 | 21 | 132
  >=65 years | 5 | 5 | 3 | 7 | 3 | 4 | 3 | 30
Age, Continuous [Median (Full Range); unit: years] | 56.0 [27 to 71] | 55.0 [25 to 73] | 53.0 [25 to 70] | 59.0 [32 to 73] | 56.0 [34 to 71] | 56.5 [21 to 72] | 53.5 [32 to 71] | 55.5 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 16 | 11 | 11 | 12 | 15 | 89
  Male | 12 | 10 | 6 | 12 | 12 | 12 | 9 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 13 | 15 | 11 | 14 | 10 | 19 | 99
  Not Hispanic or Latino | 6 | 10 | 7 | 12 | 9 | 14 | 5 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 22 | 18 | 20 | 18 | 19 | 22 | 139
  Black or African American | 1 | 0 | 3 | 3 | 3 | 2 | 0 | 12
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other (Puerto Rican) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in MRI-PDFF at Week 12 for TERN-501 Monotherapy (Arms 1, 2 and 3) Compared to Placebo.
Description: Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) is a non-invasive imaging technique that measures fat content in tissue, particularly in the liver. Relative change from baseline is calculated for each subject as 100 x [(Week 12 Value - Baseline Value)/Baseline Value].
Time Frame: 12 weeks
Population: Efficacy Analysis Set: All patients who were randomized and received at least 1 dose of the study. Primary analyses were based on observed data, i.e. no imputation was performed for missing data at Week 12. Therefore, the number of patients analyzed at Week 12 may not be the same as the number of patients treated.
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Arm 1: TERN-501 1 mg | Arm 2: TERN-501 3 mg | Arm 3: TERN-501 6 mg | Arm 7: Matching Placebo
Number analyzed (Participants) | 23 | 19 | 18 | 21
Percent change from baseline | -15.39 (5.186) | -27.48 (5.740) | -44.81 (5.856) | -4.01 (5.416)
Statistical Analysis 1: Comparison: Arm 1: TERN-501 1 mg vs Arm 7: Matching Placebo; Arm 1 compared to Placebo; Test type: Superiority; p = 0.1303, ANCOVA; Mean Difference (Final Values) = -11.39, 95% CI 2-sided [-26.178 to 3.406], Standard Error of Mean 7.480
Statistical Analysis 2: Comparison: Arm 2: TERN-501 3 mg vs Arm 7: Matching Placebo; Arm 2 compared to Placebo; Test type: Superiority; p = 0.0036, ANCOVA; Mean Difference (Final Values) = -23.47, 95% CI 2-sided [-39.140 to -7.799], Standard Error of Mean 7.924
Statistical Analysis 3: Comparison: Arm 3: TERN-501 6 mg vs Arm 7: Matching Placebo; Arm 3 compared to Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -40.80, 95% CI 2-sided [-56.545 to -25.064], Standard Error of Mean 7.960

2. Secondary Outcome: Change From Baseline in cT1 Relaxation Time at Week 12 for TERN-501 Monotherapy (Arms 1, 2 and 3) Compared to Placebo
Description: Corrected T1 (cT1) is a quantitative MRI relaxation parameter that measures liver inflammation and fibrosis. Change from baseline is calculated for each subject as (Week 12 Value - Baseline Value).
Time Frame: 12 weeks
Population: Efficacy Analysis Set: All randomized patients who received at least 1 dose of study drug. Primary analyses were based on observed data, i.e. no imputation was performed for missing data at Week 12. Therefore, the number of patients analyzed at Week 12 may not be the same as the number of patients treated.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Arm 1: TERN-501 1 mg | Arm 2: TERN-501 3 mg | Arm 3: TERN-501 6 mg | Arm 7: Matching Placebo
Number analyzed (Participants) | 22 | 19 | 18 | 21
msec | -28.2 (14.62) | -25.6 (15.71) | -72.0 (16.12) | 3.6 (14.92)
Statistical Analysis 1: Comparison: Arm 1: TERN-501 1 mg vs Arm 7: Matching Placebo; Arm 1 compared to Placebo; Test type: Superiority; p = 0.1289, ANCOVA; Mean Difference (Final Values) = -31.9, 95% CI 2-sided [-73.17 to 9.39], Standard Error of Mean 20.87
Statistical Analysis 2: Comparison: Arm 2: TERN-501 3 mg vs Arm 7: Matching Placebo; Arm 2 compared to Placebo; Test type: Superiority; p = 0.1790, ANCOVA; Mean Difference (Final Values) = -29.3, 95% CI 2-sided [-72.08 to 13.58], Standard Error of Mean 21.65
Statistical Analysis 3: Comparison: Arm 3: TERN-501 6 mg vs Arm 7: Matching Placebo; Arm 3 compared to Placebo; Test type: Superiority; p = 0.0008, ANCOVA; Mean Difference (Final Values) = -75.7, 95% CI 2-sided [-119.08 to -32.23], Standard Error of Mean 21.96

3. Secondary Outcome: Relative Change From Baseline in MRI-PDFF at Week 12 for TERN-501+TERN-101 Combination (Arms 4 and 5) Compared to Placebo
Description: as for outcome 1
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Arm 4: TERN-501 3 mg + TERN-101 10 mg | Arm 5: TERN-501 6 mg + TERN-101 10 mg | Arm 7: Matching Placebo
Number analyzed (Participants) | 19 | 21 | 21
Percent change from baseline | -20.75 (5.713) | -47.74 (5.412) | -4.01 (5.416)
Statistical Analysis 1: Comparison: Arm 4: TERN-501 3 mg + TERN-101 10 mg vs Arm 7: Matching Placebo; Arm 4 compared to Placebo; Test type: Superiority; p = 0.0358, ANCOVA; Mean Difference (Final Values) = -16.74, 95% CI 2-sided [-32.352 to -1.128], Standard Error of Mean 7.895
Statistical Analysis 2: Comparison: Arm 5: TERN-501 6 mg + TERN-101 10 mg vs Arm 7: Matching Placebo; Arm 5 compared to Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -43.73, 95% CI 2-sided [-58.858 to -28.612], Standard Error of Mean 7.647

4. Secondary Outcome: Change From Baseline in cT1 Relaxation Time at Week 12 for TERN-501+TERN-101 Combination (Arms 4 and 5) Compared to Placebo
Description: as for outcome 2
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Arm 4: TERN-501 3 mg + TERN-101 10 mg | Arm 5: TERN-501 6 mg + TERN-101 10 mg | Arm 7: Matching Placebo
Number analyzed (Participants) | 18 | 21 | 21
msec | -59.0 (16.25) | -65.5 (14.99) | 3.6 (14.92)
Statistical Analysis 1: Comparison: Arm 4: TERN-501 3 mg + TERN-101 10 mg vs Arm 7: Matching Placebo; Arm 4 compared to Placebo; Test type: Superiority; p = 0.0053, ANCOVA; Mean Difference (Final Values) = -62.6, 95% CI 2-sided [-106.33 to -18.96], Standard Error of Mean 22.09
Statistical Analysis 2: Comparison: Arm 5: TERN-501 6 mg + TERN-101 10 mg vs Arm 7: Matching Placebo; Arm 5 compared to Placebo; Test type: Superiority; p = 0.0014, ANCOVA; Mean Difference (Final Values) = -69.2, 95% CI 2-sided [-110.97 to -27.39], Standard Error of Mean 21.13

5. Secondary Outcome: Number and Percentage of Participants With Any Treatment Emergent Adverse Event for All Treatment Groups (Threshold of 0%)
Description: This outcome measures the number and percentage of participants with any Treatment Emergent Adverse Event (TEAE) for All Treatment Groups (0% Threshold). TEAEs by System Organ Class and Preferred Term meeting the 5% Threshold are reported in the Other Adverse Events section.
Time Frame: 16 weeks
Population: All 162 patients who were randomized and received at least 1 dose of study drug were included in the Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: TERN-501 1 mg | Arm 2: TERN-501 3 mg | Arm 3: TERN-501 6 mg | Arm 4: TERN-501 3 mg + TERN-101 10 mg | Arm 5: TERN-501 6 mg + TERN-101 10 mg | Arm 6:TERN-101 10 mg | Arm 7: Matching Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 24 | 24
Participants | 11 | 13 | 11 | 14 | 12 | 10 | 11

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Arm 1: TERN-501 1 mg | Arm 2: TERN-501 3 mg | Arm 3: TERN-501 6 mg | Arm 4: TERN-501 3 mg + TERN-101 10 mg | Arm 5: TERN-501 6 mg + TERN-101 10 mg | Arm 6:TERN-101 10 mg | Arm 7: Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 0/23 | 0/23 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23 | 0/22 | 0/23 | 0/23 | 2/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/23 | 8/23 | 5/22 | 10/23 | 6/23 | 5/24 | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: TERN-501 1 mg (N=23) | Arm 2: TERN-501 3 mg (N=23) | Arm 3: TERN-501 6 mg (N=22) | Arm 4: TERN-501 3 mg + TERN-101 10 mg (N=23) | Arm 5: TERN-501 6 mg + TERN-101 10 mg (N=23) | Arm 6:TERN-101 10 mg (N=24) | Arm 7: Matching Placebo (N=24)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: TERN-501 1 mg (N=23) | Arm 2: TERN-501 3 mg (N=23) | Arm 3: TERN-501 6 mg (N=22) | Arm 4: TERN-501 3 mg + TERN-101 10 mg (N=23) | Arm 5: TERN-501 6 mg + TERN-101 10 mg (N=23) | Arm 6:TERN-101 10 mg (N=24) | Arm 7: Matching Placebo (N=24)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 7 | 4 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 2 | 2 | 0 | 1 | 1
Headache (General disorders) | 1 | 1 | 1 | 2 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 3 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT05415722/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT05415722/SAP_001.pdf